CLINICAL TRIAL: NCT05283733
Title: A Prospective Randomized Controlled Trial of Reverse Conversion (Open to Laparoscopic) in Management of Acute Perforated Appendicitis
Brief Title: Open to Laparoscopic Reverse Conversion of Perforated Appendicitis
Acronym: reverse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Mohamed lotfy, Associate professor, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZUH 235
Record Dates: First submitted 2022-02-18; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Laparoscopic Surgery; Acute Appendicitis With Rupture; Sepsis; Abdominal Abscess
Keywords: laparoscopic; appendectomy; reverse conversion; reoperation; intraabdominal abscesses
MeSH Terms: conditions — Sepsis; Abdominal Abscess

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): the group who was subjected to the reverse conversion technique
  Interventions: Procedure: reverse conversion technique
- group B (No Intervention): the control group who was completed by open technique

INTERVENTIONS:
Procedure: reverse conversion technique — converting open appendectomy to laparoscopic technique for proper control of intraabdominal sepsis
  Other Names: laparoscopic lavage
  Arms: group A

SUMMARY:
A Prospective Randomized Controlled Trial of Reverse Conversion (Open to Laparoscopic) in management of Acute Perforated Appendicitis

DETAILED DESCRIPTION:
Introduction: Acute appendicitis (AA), a frequent intra-abdominal surgical pathology, necessitates a thorough awareness of its symptoms, examination, diagnosis, and total surgical management. The surgical approach to AA is appendectomy; nevertheless, the medical literature continues to argue the merits of open vs laparoscopic surgery. As with other laparoscopic surgical techniques, the literature reports lower discomfort, earlier resumption of oral feeding and shorter hospital stay following laparoscopic appendectomy (LA) as compared to open appendectomy (OA). Additionally, laparoscopy has some drawbacks such as greater cost and lengthier operating durations as compared to open surgery. The goal of this clinical study: was to compare open appendectomy versus laparoscopic conversion from open (reverse conversion) for the treatment of acute perforated appendicitis in our setting. Patients and procedures: 426 patients had perforated appendectomy and divided between two groups: group A (interventional) 213 patients who were subjected to the reverse conversion technique and group B (control)213 patients who were operated by the open technique. The key end goals for comparing both groups were the rates of intraabdominal abscess, rates of wound infection, rates of ileus and rates of reoperation. The hospital length of stay and the operative time were used as secondary end goals for comparison.

ELIGIBILITY:
Inclusion Criteria:

* symptoms consistent with acute perforated appendicitis,
* had ultrasound or computed tomography (CT) evidence of acute perforated appendicitis,
* ages ranging from 16 to 65 years.

Exclusion Criteria:

* radiological evidence of appendicular mass,
* septic shock or multi-organ failure (MOF) at presentation,
* Diabetes Mellitus (DM), renal failure, morbid obesity
* recent (6-month) history of thromboembolic disease
* immunomodulators,
* a history of inflammatory bowel disease (IBD),
* postoperative pathological report of the removed appendix revealed carcinoid or Crohn's disease,
* American Society of Anesthesiology (ASA) classification more than II.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-25 (Actual)

PRIMARY OUTCOMES:
the rates of intraabdominal abscess | 3 months post operative
  rates of complications
rates of wound infection | 3 months post operative
  rates of complications
rates of ileus | Baseline (Hospital admission)
rates of reoperation | 3 months post operative

SECONDARY OUTCOMES:
The hospital length of stay | up to 3 months
  the length of hospital stay
the operative time | Intraoperative
  Time of performing the procedures

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig University, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: Undecided